CLINICAL TRIAL: NCT05344781
Title: Relationship and Sexual Satisfaction of Stoma Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Klinikum Konstanz (Other)
Responsible Party: Principal Investigator, Silvan Haemmerli, Principal Investigator, Klinikum Konstanz
Other Study IDs: konstanz_001
Record Dates: First submitted 2021-12-07; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Satisfaction, Patient; Stoma Ileostomy; Stoma Colostomy
Keywords: Sexual satisfaction; stoma patients; relationship satisfaction
MeSH Terms: conditions — Patient Satisfaction; Orgasm | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ileostomy: Patients with ileostomy
  Interventions: Other: Questionnaire
- colostomy: Patients with colostomy
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire regarding relationship and sexual satisfaction

SUMMARY:
Anonymous questionnaire regarding relationship and sexual satisfaction as well as quality of life of stoma patients.

DETAILED DESCRIPTION:
With an anonymous questionnaire relationship, sexual and life satisfaction of stoma patients are investigated. The questionnaire will be made public by support groups and stoma nurses. Analysis of data and publication of sexual and relationship satisfaction of stoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Ileostomy or Colostomy

Exclusion Criteria:

* Disease affecting sexual functioning
* Disease affecting daily life

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ileostomy or colostomy, regardless of reason
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-20 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
sexual satisfaction | September 2022
  Questionnaire regarding sexual satisfaction of participants, multiple choice answers.
relationship satisfaction | September 2022
  Questionnaire regarding relationship satisfaction of participants, multiple choice answers.

SECONDARY OUTCOMES:
satisfaction influences | September 2022
  Questionnaire with multiple choice answers to possible influences of satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Silvan Haemmerli, Principal Investigator — Klinikum Konstanz

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT05344781/Prot_000.pdf
  • Informed Consent Form (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT05344781/ICF_001.pdf